CLINICAL TRIAL: NCT00915538
Title: A Comparison of the Bronchodilating Activity of Symbicort Pressure Metered Dose Inhaler (pMDI) 160/4.5 Used in the Conventional Manner and With a Valved Spacer Holding Chamber (Aerochamber Plus)
Brief Title: Comparing Bronchodilation of Symbicort With and Without Valved Holding Chamber (Aerochamber Plus)
Acronym: WSMR2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Western Sky Medical Research (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Lyndon Mansfield, Director, Western Sky Medical Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: WSMR 2008-2
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Asthma
Keywords: Asthma; Formoterol; Long Acting Beta Adrenergic Bronchodilator; Symbicort; Aerochamber
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 / use of pMDI as approved (Other): The intervention in this group will use inhalation from the pMDI containing budesonide/formoterol pMDI 160/4.5 2 inhalations as approved. (FDA approved product information) without a spacer. The pulmonary function tests (PFTs) will be collected at baseline and for a period of 12 hours post inhalation of 2 inhalation of budesonide /formoterol; pMDI160/5.
  Interventions: Drug: pMDI budesonide/formotrol 160/4.5 is in group 1; Device: Symbicort 160/4.5 plus Aerochamber Plus included in group 2
- Group 2 / pMDI with Aerochamber Plus (Experimental): The intervention in this group will use the pMDI budesonide/formoterol 160/4.5 with a valve holding chamber spacer device, Aerochamber Plus which is the intervention being studied The PFTs will be collected at baseline and for a period of 12 hours post inhalation of 2 inhalation of Symbicort 160/5. This is the intervention to be studied for comparison to the non-spacer inhalations..
  Interventions: Drug: pMDI budesonide/formotrol 160/4.5 is in group 1; Device: Symbicort 160/4.5 plus Aerochamber Plus included in group 2

INTERVENTIONS:
Drug: pMDI budesonide/formotrol 160/4.5 is in group 1 — The asthmatic subjects will receive budesonide/formoterol pMDI 160/4.5 pMDI 2 inhalations used in conventional fashion, and have pulmonary function measured over 12 hours who are expected to show bronchodilation.
  Other Names: Symbicort
Device: Symbicort 160/4.5 plus Aerochamber Plus included in group 2 — Symbicort 160/4.5 2 inhalations will be administered through a valved holding chamber, Aerochamber Plus, Pulmonary functions will be measured over 12 hours in asthmatic subjects who are expected to show bronchodilation.
  Other Names: Symbicort; Aerochamber plus

SUMMARY:
This study will compare the amount of bronchial tube relaxation from the Formoterol medicine contained in the Symbicort pressure Metered Dose Inhaler(pMDI)(a combination of Budesonide, a steroid, and Formoterol, a drug which relaxes the bronchial smooth muscle. The comparison will be using the pMDI in the usual fashion to the pMDIs and a spacer which allows more time for breathing in the medication. Breathing tests will be measured over a 12 hour period for the comparison.

DETAILED DESCRIPTION:
Sixteen subjects will receive treatment in a cross-over design. They will inhale Symbicort 160/4.5 two inhalations in the manner prescribed in the approved package insert. The second intervention will be the inhalation of Symbicort 160/4.5 two inhalations through a valved holding chamber (Aero Chamber Plus). Breathing tests including spirometry will be measured at various time periods over a 12-hour time frame in each intervention. Comparison will be made of the two periods to demonstrate that the use of the valved holding chamber does not adversely affect the bronchodilation of the formoterol component of the combination drug.

ELIGIBILITY:
Inclusion Criteria:

* Asthma with 15% or more increase in Forced expiratory volume at 1 second (FEV-1) after 180-360 mcg of albuterol pMDI

Exclusion Criteria:

* Any illness or condition which might place subject at risk in the study;e.g. some cardiovascular disorders Inability to understand and sign informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon E Mansfield, MD, Principal Investigator — Western Sky Medical Research
Locations (1):
- Western Sky Medical Research, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The results were published in the Journal of Asthma . 2013 Feb :50(1)71-4. Dr. Mansfield was the corresponding author and could be reached by email or phone regarding the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: February 2013
Access Criteria: Query to the corresponding author

REFERENCES:
- [Background] Dolovich MB, Ahrens RC, Hess DR, Anderson P, Dhand R, Rau JL, Smaldone GC, Guyatt G; American College of Chest Physicians; American College of Asthma, Allergy, and Immunology. Device selection and outcomes of aerosol therapy: Evidence-based guidelines: American College of Chest Physicians/American College of Asthma, Allergy, and Immunology. Chest. 2005 Jan;127(1):335-71. doi: 10.1378/chest.127.1.335. PMID 15654001
- [Background] Newman SP. Principles of metered-dose inhaler design. Respir Care. 2005 Sep;50(9):1177-90. PMID 16122401
- [Background] Hess DR. Aerosol delivery devices in the treatment of asthma. Respir Care. 2008 Jun;53(6):699-723; discussion 723-5. PMID 18501026
- [Derived] Mansfield LE, Maynes R. A valved holding chamber does not decrease the bronchodilator activity of budesonide-formoterol combination metered dose inhaler. J Asthma. 2013 Feb;50(1):71-4. doi: 10.3109/02770903.2012.745093. Epub 2012 Nov 26. PMID 23176189

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional First: This group will use pMDI in usual fashion first and cross over to pMDI and valved holding chamber
- Spacer First: This arm will receive pMDI and Valved holding chamber on fist day. On anther day will receive pMDI in usual fashion. Pulmonary functions wil be measured over 12 hours
Period: Overall Study
Arm/Group | Conventional First | Spacer First
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional First | Spacer First | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (7) | 36 (7) | 36.5 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Mean Area Under the Curve (AUC) of Forced Expiratory Volume in One Second (FEV-1) Over 12 Hours, Measured (BL), 5, 10, 15, 60, 120, 240, 480, 720 Minutes. The Unit is Liters, and the AUC is in Liters.
Description: The mean FEV-1 (Forced Expiratory Volume 1 second) for each of the treatments (with and without valved holding chamber) in this crossover design were recorded at BL, 5, 10, 15, 30, 60, 120, 240. 480, 720 minutes (12 hrs) were plotted as a curve and the area under the curve was calculated. The measured results was mean liters/12 hours.
Time Frame: BL, 5, 10,15,30,60,120,240,480,720 minutes (12 hrs)
Measure: Mean (Full Range); unit: Liters X hours
Groups:
- Group 1: The intervention in this group will inhalation from the pMDI containing budesonide/formoterol pMDI 160/4,5 2 inhalations as recommended in product PI (FDA approved product information)without a spacer. The pulmonary function tests (PFTs) will be collected at baseline and for a period of 12 hours post inhalation of 2 inhalation of budesonide /formoterol; pMDI160/5.
  pMDI budesonide/formotrol 160/4.5 is in group 1: The subjects will receive budesonide/formoterol pMDI 160/4.5 pMDI used in conventional fashion, and have pulmonary function measured over 12 hours.
  Symbicort 160/4.5 plus Aerochamber Plus icluded in group 2: Symbicort 160/4.5 will be administered through a valved holding chamber, Pulmonary functions will be measured over 12 hours.
- Group 2: The intervention in this group will use the pMDI budesonide/formoterol 160/4.5 with a valve holding chamber spacer device (aerochamber plus)which is the intervention being studied The PFTs will be collected at baseline and for a period of 12 hours post inhalation of 2 inhalation of Symbicort 160/5. This is the intervention to be studied for comparison to the non-spacer inhalations..
  pMDI budesonide/formotrol 160/4.5 is in group 1: The subjects will receive budesonide/formoterol pMDI 160/4.5 pMDI used in conventional fashion, and have pulmonary function measured over 12 hours.
  Symbicort 160/4.5 plus Aerochamber Plus icluded in group 2: Symbicort 160/4.5 will be administered through a valved holding chamber, Pulmonary functions will be measured over 12 hours.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 16 | 16
Liters X hours | 2.77 [0 to 720] | 2.79 [0 to 720]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; The cross-over means there were 16 determinants for each time for each treatment. The AUC of FEV-1 was measured in each subject for each treatment arm and the mean of this data was compared; Test type: Non-Inferiority or Equivalence — The expected results for non-inferiority would be +/- 5% of difference between the two groups in the primary efficacy parameter; p = 0.76, t-test, 2 sided; AUC = 0.0
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Test type: Other — Two sample T test; p > .05, t-test, 2 sided; Mean Difference (Net) = 0, Standard Deviation 12

2. Secondary Outcome: FEV-1/FVC
Description: The ratio of the volumes in liters of FEV-1 to Forced vital capacity (FVC). This is reported as percent for each time point., Each time point will be compared.for the two interventions. This expressed as a percentage.
Time Frame: 0,5,10,15,30,60,120,240,480,720 minutes
Population: This is a cross over design. 2 cohorts of 8 subjects will be tested in a cross over design, so that 16 measurements will be made for each intervention. This should give power of 0.8 for non inferiority equivalence study.
Measure: Mean (Standard Deviation); unit: percentage of fev1/fvc
Groups:
- Spacer: This arm will receive pMDI Symbicort 160/4.5 with an Aerochamber Plus Valved holding chamber.
- Non-Spacer (Conventional): This arm will receive pMDI Symbicort 160/4.5 without an Aerochamber.
Arm/Group | Spacer | Non-Spacer (Conventional)
Number analyzed (Participants) | 16 | 16
percentage of fev1/fvc
  0 time | 76.13 (11.7) | 75.58 (12.5)
  5 minutes | 79.08 (12.07) | 79.91 (14.33)
  10 minutes | 78.55 (13.53) | 81.16 (15.08)
  15 minutes | 79.08 (10.80) | 80.29 (13.13)
  30 minutes | 80.17 (14.32) | 80.55 (15.11)
  60 minutes | 78.05 (15.30) | 81.63 (14.63)
  120 minutes | 80.94 (13.95) | 81.40 (15.97)
  240 minutes | 81.56 (14.30) | 82.42 (13.75)
  480 minutes | 79.95 (14.43) | 80.56 (13.94)
  720 minutes | 79.93 (12.54) | 80.33 (13.36)
Statistical Analysis 1: Comparison: Spacer; The cross over means there were 16 determinants for each time for each treatment; Test type: Non-Inferiority or Equivalence — Power calculation was not done for secondary parameter. The comparison was for the FEV-1/FVC expressed as fraction at each time point; p = 0.76, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected during a period of two weeks (the study duration).
Description: No source vocabulary was used as there were no adverse events to record. No table was formed because of no data.
Groups:
- Conventional: This group will use pMDI in usual fashion
- Spacer: This arm will receive pMDI and Valved holding chamber
Arm/Group | Conventional | Spacer
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
No subject discontinued subjects were adults experienced in using a pressured metered dose inhaler (pMDI), Spacers or holding chambers are most frequently used by patients with coordination difficulties.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No